CLINICAL TRIAL: NCT05606055
Title: Phase IV, Single-center, Open Study to Evaluate the Benefits of the Start of Immediate Treatment Without Immunovirological Data ("Same Day Treatment") Compared to Conventional Treatment With BIC / FTC / TAF (Bictegravir/Emtricitabina/Tenofovir) in Naive Patients With Type 1 HIV (Human Immunodeficiency Virus) Infection
Brief Title: The Benefits of Immediate Treatment Initiation Without Immunovirological Data Compared to Conventional BIC / FTC / TAF Treatment in Naive Patients With Type 1 HIV (Human Immunodeficiency Virus) Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, Irene Carrillo, Subinvestigator Infectious disease. Irene Carrillo, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2022-09-15; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDT (Experimental): -75 patients of immediate treatment, will be those patients without immuno-virological data that accept to start the treatment the same day of the first consultation with the hospital specialist (arm 1 or SDT).
  Interventions: Drug: BIC/FTC/TAF: Bictegravir/emtricitabina/tenofovir alafenamida fumarato
- Conventional (Active Comparator): - 75 patients of conventional treatment, will be those who in their first consultation with the hospital specialist already have previous immuno-virological data or reject the start of immediate treatment (arm 2 or conventional).
  Interventions: Drug: BIC/FTC/TAF: Bictegravir/emtricitabina/tenofovir alafenamida fumarato

INTERVENTIONS:
Drug: BIC/FTC/TAF: Bictegravir/emtricitabina/tenofovir alafenamida fumarato — This is a study to assess the impact of immediate ART (FAST ART or SDT) against conventional treatment (CT) on the time to reach an undetectable HIV-1 viral load.

SUMMARY:
Phase IV, single-center, open study to assess the benefits of the start of immediate treatment without immunovirological data ("Same Day Treatment") compared to conventional treatment with BIC / FTC / TAF in naive patients with type 1 HIV (human immunodeficiency virus) infection

DETAILED DESCRIPTION:
150 patients (75 in each treatment arm) with a confirmed diagnosis of HIV-1 infection and without prior antiretroviral treatment will be included.

Expected study period 48 weeks of treatment Main objective of effectiveness Determine the time from the first determination of CD4 and HIV-1 viral load to achieve HIV viral load <50 cop / ml.

Secondary objectives of efficacy

* Evaluate changes in CD4 T cell count.
* Determine the time from HIV diagnosis to achieve undetectable HIV viral load.
* Determine the degree of anxiety of patients.
* Determine the number of sexual contacts with potential for transmission of HIV infection.
* Determine the quality of patients before and after SDT. Both arms of the study have the same treatment with triple therapy (BIC / FTC / TAF).

The treatment guidelines will be as follows:

* Patients in the immediate treatment arm (SDT) will take 1 tablet (50 mg BIC + 200 mg FTC + 25 mg TAF) orally, once a day, from the moment they are seen in the specialist's office (without immunovirological data information).
* Patients in the conventional treatment arm will take 1 tablet (50 mg BIC + 200 mg FTC + 25 mg TAF) orally, once a day, from the moment the immunovirological results are obtained (either because it is available them at the first visit with the specialist, or because the patient wishes to wait for such information prior to the start of the treatment).

It is a single-center, open and non-randomized study. 150 adult patients with confirmed diagnosis of HIV-1 and without prior antiretroviral treatment may participate in the study.

Patients will be divided into two groups, one in immediate treatment (arm 1 or SDT) and another in conventional treatment (arm 2), both strategies being considered part of the usual clinical practice that leads to a low intervention study.

* 75 patients of immediate treatment, will be those patients without immuno-virological data that accept to start the treatment the same day of the first consultation with the hospital specialist (arm 1 or SDT).
* 75 patients of conventional treatment, will be those who in their first consultation with the hospital specialist already have previous immuno-virological data or reject the start of immediate treatment (arm 2).

Patients will voluntarily grant informed consent before performing any study procedure and will be assigned a patient code for the entire study.

The study will include a total of 5 visits and periodic clinical exams will be performed on visits of weeks 0, 4, 12, 24 and 48.

ELIGIBILITY:
Inclusion Criteria:

- Men and women > 18 years old

* Confirmed and documented diagnosis of HIV-1 infection
* Without prior antiretroviral treatment (excluding 28-day post-exposure prophylaxis)
* Signed informed consent
* Negative pregnancy test (women of childbearing age only). Women of childbearing age are considered to be those women who have not undergone permanent infertility procedures or who have been amenorrheic for less than 12 months

Exclusion Criteria:

* Inability to obtain written informed consent to participate in the study
* Pregnant or breastfeeding women or those who intend to become pregnant during the study period and do not undertake to use proven contraceptive methods
* Any suspicion or confirmation of resistance to TAF, FTC or BIC
* Estimated glomerular filtration rate (TFGe) <30 mg / ml / m2 measured by any of the available formulas. The determination of the TFGe of a routine prior analysis of ≤ 12 weeks prior to the signing of the consent is allowed
* Contraindications to the use of TAF
* Clinical condition of the patient in rapid deterioration or the investigator considers that there is no reasonable hope that the patient will end the study
* Simultaneous participation in another clinical trial or research study that requires the need for treatment with other drugs outside the study or interferes with visits to it.
* Any situation that, in the opinion of the investigator, may interfere with the patient's ability to comply with the treatment schedule and protocol evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of immediate treatment. | 48 weeks
  The time in weeks from the first determination of CD4 and HIV-1 viral load until achieving HIV viral load <50 cop/ml, in number.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoints | 48 weeks
  * CD4 cell count in number
  * Time from HIV diagnosis to achieving undetectable HIV viral load, in weeks.
  * Degree of anxiety of patients (mild, moderate and severe degree according to the HADS scale).
  * Number of sexual contacts with potential for transmission of HIV infection, in number.
  * Quality of patients before and after SDT, según escala EQ-5D 5 (numerical value from 1 to 5).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital FUNDACIÓN JIMÉNEZ DÍAZ, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marks G, Crepaz N, Janssen RS. Estimating sexual transmission of HIV from persons aware and unaware that they are infected with the virus in the USA. AIDS. 2006 Jun 26;20(10):1447-50. doi: 10.1097/01.aids.0000233579.79714.8d. PMID 16791020
- [Result] Gallant J, Lazzarin A, Mills A, Orkin C, Podzamczer D, Tebas P, Girard PM, Brar I, Daar ES, Wohl D, Rockstroh J, Wei X, Custodio J, White K, Martin H, Cheng A, Quirk E. Bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir, abacavir, and lamivudine for initial treatment of HIV-1 infection (GS-US-380-1489): a double-blind, multicentre, phase 3, randomised controlled non-inferiority trial. Lancet. 2017 Nov 4;390(10107):2063-2072. doi: 10.1016/S0140-6736(17)32299-7. Epub 2017 Aug 31. PMID 28867497
- See also: UNAIDS is leading the global effort to end AIDS as a public health threat by 2030 as part of the Sustainable Development Goals. — https://www.unaids.org/en
- See also: GUIDELINES FOR MANAGING ADVANCED HIV DISEASE AND RAPID INITIATION OF ANTIRETROVIRAL THERAPY — https://apps.who.int/iris/bitstream/handle/10665/255884/9789241550062-eng.pdf;jsessionid=BB91240E0947C3461F781F6FBC9E3B49?sequence=1